CLINICAL TRIAL: NCT01851876
Title: Endometrial Injury May Increase the Clinical Pregnancy Rate in Normoresponders Underwent Long Agonist Protocol Intracytoplasmic Sperm Injection Cycles With Single Embryo Transfer
Brief Title: Endometrial Injury and Single Embryo Transfer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Suleyman Guven, Assoc. Prof., Karadeniz Technical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011/20
Record Dates: First submitted 2013-04-26; First posted 2013-05-13 (Estimated); Results first posted 2013-07-01 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2013-05

CONDITIONS: Primary Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endometrial injury (Experimental): The patients in this group will be subjected to endometrial injury procedure in preceding IVF cycle.
  Interventions: Device: Endometrial injury
- No endometrial injury (No Intervention): The patients in this group will not be subjected to endometrial injury procedure in presiding IVF cycle. The patients will be stimulated with standard IVF protocol.

INTERVENTIONS:
Device: Endometrial injury — Endometrial injury with Endometrial Suction Curette (pipelle) will be performed.
  Arms: Endometrial injury

SUMMARY:
Endometrial injury increases clinical pregnancy rate in normoresponder patients undergoing long agonist protocol intracytoplasmic sperm injection cycles with single embryo transfer.

DETAILED DESCRIPTION:
Endometrial injury means endometrial biopsy on day 3 of menstrual cycle following down regulation in an IVF patient.

ELIGIBILITY:
Inclusion Criteria:

* woman age under 35 years
* history of primary infertility
* normoresponder (antral follicle count 5-10 in one ovary in early follicular phase
* having grade I or II embryos for transfer
* agree to undergo endometrial biopsy during the COH cycle. All patients were stimulated with luteal phase long protocol.

Exclusion Criteria:

* endocrinopathies (including diabetes mellitus, hyperprolactinemia, Cushing's disease, and congenital adrenal hyperplasia), any systemic disease, collagen disorder, hypercholesterolemia, sickle cell anemia, and a history of neoplasm; -high risk for or history of OHSS
* using any concurrent medication (e.g., insulin-sensitizing drugs, and GnRH antagonists)
* patients who did not proceed to follicle retrieval
* severe male infertility requiring TESA/TESA
* mullerian tract anomalies
* a history of endometrial instrumentation or surgery within a month of the study
* not agree to undergo endometrial biopsy during the COH cycle.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2010-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suleyman Guven, Principal Investigator — Karadeniz Technical University

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One hundred thirty consecutive women undergoing 130 ICSI cycles between September 2010 to April 2011 at our clinic were included for this prospective case control study.
Pre-assignment Details: Following inclusion/exlusion criteria 9 women were excluded for study group, while 5 women for control group.
Period: Overall Study
Arm/Group | Endometrial Injury | No Endometrial Injury
Started | 56 | 62
Completed | 56 | 62
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Endometrial Injury | No Endometrial Injury | Total
Number analyzed (Participants) | 56 | 62 | 118
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 56 | 62 | 118
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 30.83 (2.90) | 31.14 (2.95) | 31.0 (2.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 62 | 118
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Turkey | 56 | 62 | 118

OUTCOME MEASURES:

1. Primary Outcome: Clinical Pregnancy Rate
Time Frame: up to 6 months
Reporting Status: Not Posted

2. Primary Outcome: Clinical Pregnancy Rate
Time Frame: 4 months
Measure: Number; unit: participants
Arm/Group | Endometrial Injury | No Endometrial Injury
Number analyzed (Participants) | 56 | 62
participants | 27 | 18
Statistical Analysis 1: Comparison: Endometrial Injury vs No Endometrial Injury; Test type: Superiority or Other; p = 0.025, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Endometrial Injury | No Endometrial Injury
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
No limitations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes